CLINICAL TRIAL: NCT02742350
Title: Effects of Inspiratory Muscle Training Hihg Intensity Linked to Cardiac Rehabilitation in Patients on Exercise Performance in the Post-operative of Coronary Artery Bypasssurgery: a Randomized Clinical Trial
Brief Title: Effects of Muscle Trainins Inspiratory Linked to Cardiac Rehabilitation Post-operative of CABG Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Clinical Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMT+exercise-CABG
Record Dates: First submitted 2016-03-07; First posted 2016-04-19 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT+Exercise (Experimental): The inspiratory muscle training protocol (IMT) high intensity is achieved with a device with linear load pressure (POWERbreathe Plus Light Resistance®, SP, BR) that allows loads up to -90cmH2O. IMT is performed for 36 sessions (12 weeks) with weekly frequency of three times a week under supervision prior to the cardiac rehabilitation. The training protocol consists of five series with 10 repetitions each set until the 8th week with increase in the number of sets of repetitions of the 8th to 12th week, with two minutes or according to patient feedback using the modified Borg scale . Aerobic training lasts 40 minutes (5 minutes heating 30 minute workout and 5 minutes desaqueciemento. During training vital signs such as heart rate, blood pressure (BP) and peripheral oxygen saturation (SpO2) are evaluated and the feeling of effort the patient should not exceed the level of 8 according to the modified Borg scale.
  Interventions: Device: IMT - POWERbreathe Plus Light Resistance®, SP, BR
- Exercise Control (No Intervention): Aerobic Exercise and Stretching

INTERVENTIONS:
Device: IMT - POWERbreathe Plus Light Resistance®, SP, BR — POWERbreathe Plus Light Resistance®, SP, BR
  Arms: IMT+Exercise

SUMMARY:
Heart surgery procedures are still widely used worldwide for the treatment of patients with heart problems, and rates of complications in the postoperative period related to them remain high. In these patients, physical conditioning programs result in improved functional capacity, and reducing the heart rate and systolic blood pressure. The inspiratory muscle training is also emerging as a valuable strategy in the treatment of cardiac patients. The study of the interaction between cardiac rehabilitation and high intensity IMT about these changes is not yet understood in this population. The aim of this study is to assess the effects of inspiratory muscle training high intensity associated with cardiac rehabilitation exercise performance of patients in the postoperative period of CABG surgery.

DETAILED DESCRIPTION:
It is a controlled, randomized clinical trial in which patients were randomly assigned randomly after referral to cardiac rehabilitation: Group 1 IMT-HI, group 2 - IMT-HI control. The evaluator of outcomes is blinded as to groups. The study protocol lasts 36 sessions for both groups. The group 1 patients performs cardiac rehabilitation protocol for 40 minutes with cardio and stretching and also inspiratory muscle training protocol of high intensity with 50% load increase in maximal inspiratory pressure during the first two weeks, 60% of MIP in third and fourth week, 70% of MIP in the fifth and sixth week and 80% MIP in the seventh and eighth week. The group 2 patients only perform the cardiac rehabilitation protocol for 40 minutes with aerobic exercise and stretching.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the postoperative period of elective CABG
* Between the fourteenth and the thirtieth day after surgery
* Between 30 and 70 years old

Exclusion Criteria:

* Decompensated heart failure
* Unstable angina
* Moderate respiratory disease severe
* Active infectious disease or fever
* Disabling peripheral vascular disease
* Unstable ventricular arrhythmias
* Use of cardiac pacemaker.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | 1 week, up to 4 week, up to 8 week, through study completion, an average of 12 week
  The patient is set to walk in a corridor of 30 meters delimited cones for six minutes in order to go as far as possible. Every minute the patient is stimulated by the evaluator.

SECONDARY OUTCOMES:
30-s chair-stand | 1 week, up to 4 week, up to 8 week, through study completion, an average of 12 week
  With the patient sitting in a chair with 45cm tall, with your feet apart and flat on the floor and arms crossed against his chest, the patient will be encouraged to get up and return to a sitting position as many times as possible in 30 seconds, It is registered the maximum number of repetitions.
respiratory muscle strength test | 1 week, up to 4 week, up to 8 week, through study completion, an average of 12 week
Quality of life | 1 week, through study completion, an average of 12 week
  Brazilian version of the Quality of Life Questionnaire - SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Della Méa Plentz, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No